CLINICAL TRIAL: NCT04973644
Title: Combining Wearable Technology to Crate Internet+Digital Hospital-remote Home Type 2 Diabetes Follow-up Management Mode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, YunFeng Shen, professor, Second Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM202106
Record Dates: First submitted 2021-07-07; First posted 2021-07-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet + Digital Hospital-remote home management mode (Experimental): Remote monitoring devices+Internet management platform, dietary recommendations, exercise supervision, web education, information pushing, doctor-patient interaction.
  Interventions: Device: Remote monitoring devices+Internet management platform
- the traditional management mode (No Intervention): Routine dietary and exercise recommendations, education as well as monitor in the clinic.

INTERVENTIONS:
Device: Remote monitoring devices+Internet management platform — Remote monitoring devices collects blood glucose, total cholesterol, serum ketones and serum uric acid,then upload data to the platform.
  Arms: Internet + Digital Hospital-remote home management mode

SUMMARY:
This study intends to combining wearable technology to crate Internet+Digital Hospital-remote Home Type 2 Diabetes follow-up management mode.To preliminarily explore compared with the traditional medical treatment mode, whether the new management mode of DM can improve the management objectives and patient satisfaction of T2DM and reduce medical costs. The study provides a powerful reference for establishing corresponding platforms and promoting such models at the government management level in the future.

DETAILED DESCRIPTION:
Background:The prevalence of T2DM in Chinese adults has exceeded 10%, and the prevalence of abnormal glucose metabolism has exceeded 40% in people older than 18 years. This will lead to a significant increase in the prevalence of DM complications in the next decade, and the disability and death caused by complications will also seriously affect the quality of life of patients and bring a huge social and economic burden.This randomized controlled trial intends to combining wearable technology to crate Internet+Digital Hospital-remote Home T2DM follow-up management mode.To preliminarily explore compared with the traditional medical treatment mode, whether the new management mode of DM can improve the management objectives and patient satisfaction of T2DM and reduce medical costs. The study provides a powerful reference for establishing corresponding platforms and promoting such models at the government management level in the future.

Methods:The study was a parallel-group, randomised, controlled trial. the number of cases planned to be included in 200 cases. Participants were randomly assigned to the intervention or control group.The intervention group receives Internet + Digital Hospital-remote home management mode,including remote monitoring devices+Internet management platform, dietary recommendations, exercise supervision, web education, information pushing, doctor-patient interaction, etc.The control group receives the traditional management mode, including routine dietary and exercise recommendations, education as well as monitor in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes according to the World Health Organization criteria;
* Aged between 18 and 70 years;
* Glycosylated haemoglobin (HbA1C%) between 7% and 9%.

Exclusion Criteria:

* Type 1 diabetes;
* Gestational diabetes;
* Other special types of diabetes;
* Moderate-severe insufficiency of heart , liver, kidney and lung;
* Complicated with acute disease or stress status.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-08-21 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-07-23 (Actual)

PRIMARY OUTCOMES:
HbA1c concentration | Baseline, Week 12, Week 24
  HbA1c concentration reflects the average blood glucose level

SECONDARY OUTCOMES:
FBG | Baseline, Week 24
  Normal FBG values are 3.9 to 6.1 mmol/L
Fasting insulin | Baseline, Week 24
  Insufficient insulin secretion or insulin resistance is a major cause of diabetes
Blood pressure | Baseline, Week 24
  Normal systolic blood pressure <140mm Hg, diastolic blood pressure<90mmHg in China.
Total cholesterol | Baseline, Week 24
  Total cholesterol refers to the sum of cholesterol contained by all lipoproteins in the blood.Normal Total cholesterol values <5.17 mmol/L
Triglycerides | Baseline, Week 24
  Normal Triglycerides values Triglycerides<1.7 mmol/L
LDL-C | Baseline, Week 24
  The level of LDL-C is correlated with the incidence and severity of cardiovascular disease
HDL-C | Baseline, Week 24
  The level of HDL-C is inversely associated with coronary heart disease.
Weight | Baseline, Week 24
  Standard weight is one of the important signs to reflect and measure a person's health status
Waist circumference | Baseline, Week 24
  Waist circumference is an important index to determine central obesity.
BMI | Baseline, Week 24
  BMI is an internationally used measure of how fat and thin a person is and whether they are healthy or not.The calculation formula is: BMI= weight/height^2.
Serum uric acid | Baseline, Week 24
  Serum uric acid is the end product of purine catabolism.Is excreted by the kidney with urine.Serum uric acid measurement is a sensitive marker for the diagnosis of severe renal impairment.
Serum creatinine | Baseline, Week 24
  Clinically detecting serum creatinine is one of the main methods to understand renal function, and it is an important indicator of kidney function, and an elevated serum creatinine means the damage of kidney function.
Urinary microalbumin / creatinine ratio | Baseline, Week 24
  Urinary microalbumin /creatinine ratio is the test used clinically to judge microalbuminuria, examine early renal lesions, and is more commonly used clinically for early diabetic nephropathy.
Diabetes Treatment Satisfaction Questionnaire | Week 24
  Comments on the distribution of treatment satisfaction scores measured by the Diabetes Treatment Satisfaction Questionnaire (DTSQ).There are 8 items in total, including three dimensions of treatment satisfaction, self-perceived hyperglycemia and self-perceived hypoglycemia.The minimum and maximum values are 0 and 36 ,respectively.Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi, China

REFERENCES:
- [Derived] Peng P, Shen Y, Xiong H. Wearable monitoring device based on an internet management platform improves metabolic parameters in type 2 diabetes patients: a prospective pilot study. Postgrad Med. 2024 Jun;136(5):523-532. doi: 10.1080/00325481.2024.2366156. Epub 2024 Jun 13. PMID 38870076